CLINICAL TRIAL: NCT02288754
Title: Detection of Tumor DNA in Blood Samples From Patients With Late Stage Cancer and "Healthy Controls"
Brief Title: Detection of Tumor DNA in Blood Samples From Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lexent Bio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LB1985106
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Cancer; Tumors
Keywords: DNA in Tumors; cfDNA; WGS; Advanced stage cancer; Solid tumors
MeSH Terms: conditions — Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood 2 x 10 ml of Streck; FFPE tumor tissue (optional)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stage II or III curative surgery (closed to accrual): Patients with stage II or III solid tumors undergoing curative intend surgery enrolled before surgery.
  Interventions: Diagnostic Test: Blood test
- Stage II or III neoadjuvant therapy cohort (closed to accrual): Patients with stage II or III solid tumors undergoing neoadjuvant therapy followed by curative intend surgery enrolled before neoadjuvant therapy.
  Interventions: Diagnostic Test: Blood test
- Metastatic disease: Patients with advanced, recurrent and/or metastatic disease requiring systemic therapy with chemotherapy, targeted therapy, immunotherapy or a combination of any before initiation of any therapy or a new line of therapy following documentation of disease progression on prior therapy.
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — No intervention except to collect blood for diagnostic test development

SUMMARY:
The aim of this study is to employ genomic detection methodologies to measure the relative amount of tumor nucleic acids in the blood of a cancer patient with diagnosed metastatic disease that is either commencing, currently undergoing or completed cytotoxic chemotherapy treatment. More generally, this approach will allow us to develop a quantitative measure of therapy efficacy via the counting of the relative changes in tumor molecules over the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Have metastatic disease with from a solid tumor (e.g. breast, lung, colon, pancreas, ovary, prostate...) or stage II or III solid tumors undergoing curative surgery or neoadjuvant therapy followed by surgery
* Starting treatment or a new line of treatment
* Able to understand and grant informed consent
* Able to have their blood drawn

Exclusion Criteria:

* Unable to grant informed consent or comply with all study procedures.
* Has a hematological malignancy, i.e. myeloma, lymphoma, MDS, leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are (i) commencing or (ii) starting a new line of treatment for metastatic disease with any cytotoxic chemotherapy, targeted therapy, immunotherapy, a combination of any and/or radiation therapy. Patients with stage II or III solid tumors undergoing curative intend surgery or neoadjuvant therapy followed by surgery are also eligible, before surgery or initiation of neoadjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-12; Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Correlation between the tumor load score and patient response to therapies. | 5 years
  Determination of a direct correlation between the tumor load score and patient response to therapies.

SECONDARY OUTCOMES:
Determination of particular mutation events which underlie the basis of any established correlation with therapy response. | 5 years
  To determine which particular mutation events underlie the basis of any established correlation with therapy response.

CONTACTS AND LOCATIONS:
Overall Officials: Haluk Tezcan, MD, Principal Investigator — Lexent Bio
Locations (1):
- Cancer Care Associates, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No